CLINICAL TRIAL: NCT02298543
Title: The Multicenter Registry to Evaluate the Natural Course of Coronary Spasm Patients Presenting Aborted Sudden Cardiac Death
Brief Title: Coronary Spasm Presenting Aborted Sudden Cardiac Death, the Multicenter Registry
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-11
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Vasospasm; Cardiac Death
MeSH Terms: conditions — Coronary Vasospasm; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary spasm
  Interventions: Other: coronary spasm

INTERVENTIONS:
Other: coronary spasm

SUMMARY:
The purpose of this study is to evaluate the natural course of coronary spasm patients presenting aborted sudden cardiac death and analyze risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Coronary spasm

Exclusion Criteria:

* Life expectancy less than 2years
* Coronary stenosis 50% and more
* Structural abnormalities of the heart leading to ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary spasm
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
all cause death | 1 year
myocardial infarction | 1 year
ventricular tachycardia | 1 year
ventricular Fibrillation | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea